CLINICAL TRIAL: NCT02612922
Title: A Phase III Randomized Double-Blind Placebo Controlled Trial to Evaluate the Efficacy and Safety of Nitazoxanide in the Treatment of Acute Uncomplicated Influenza
Brief Title: Trial to Evaluate the Efficacy and Safety of Nitazoxanide in the Treatment of Acute Uncomplicated Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM08-3003
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitazoxanide (Active Comparator): Two Nitazoxanide 300 mg tablets orally twice daily (b.i.d.) for 5 days
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): Two Placebo tablets orally twice daily (b.i.d.) for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide 600 mg administered orally twice daily for five days
  Other Names: NTZ, Alinia
  Arms: Nitazoxanide
Drug: Placebo — Placebo administered orally twice daily for five days
  Arms: Placebo

SUMMARY:
Trial to evaluate efficacy and safety of nitazoxanide (NTZ) in the treatment of acute uncomplicated influenza.

DETAILED DESCRIPTION:
A multicenter randomized double-blind placebo controlled trial designed to evaluate efficacy and safety of NTZ 600 mg administered orally twice daily for five days compared to a placebo in the treatment of acute uncomplicated influenza.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 to 65 years
2. Presence of clinical signs and/or symptoms consistent with an acute illness compatible with influenza infection (each of the following is required):

   * oral temperature of ≥100.4°F or ≥38°C (obtained in office or self-measured within 12 hours prior to screening - if self-measured, subject must also have taken an antipyretic within 4 hours prior to screening) AND
   * at least one of the following respiratory symptoms (cough, sore throat, nasal obstruction), AND
   * one of the following constitutional symptoms (fatigue, headache, myalgia, feverishness).
3. Confirmation of influenza A or B infection in the local community by one of the following means:

   * the institution's local laboratory,
   * the local public health system,
   * the national public health system, or
   * a laboratory of a recognized national or multinational influenza surveillance scheme.
4. Onset of illness no more than 40 hours before enrollment in the trial.

   Note: Time of onset of illness is defined as either the earlier of:
   * the time when the temperature was first measured as elevated, OR
   * the time when the subject experienced the presence of at least one respiratory symptom AND the presence of at least one constitutional symptom.
5. Willing and able to provide written informed consent (including assent by legal guardian if under 18 years of age) and comply with the requirements of the protocol, including completion of the patient diary.

Exclusion Criteria:

1. Severity of illness requiring or anticipated to require in-hospital care or subject defined as being at high risk of complications from influenza infection according to the Infectious Diseases Society of America (IDSA) guidelines for seasonal influenza in adults and children (Committee of Infectious Diseases (CID) 2009:48) or current Centers for Disease Control and Prevention (CDC) criteria. Current criteria for persons 12-65 years of age who are at risk of influenza complications include (list to be reviewed and updated as required prior to initiation of the study and at least monthly during the study):

   * Persons with asthma or other chronic pulmonary diseases, such as cystic fibrosis in children or chronic obstructive pulmonary disease in adults.
   * Persons with hemodynamically significant cardiac disease.
   * Persons who have immunosuppressive disorders or who are receiving immunosuppressive therapy.
   * Human Immunodeficiency Virus (HIV) infected persons.
   * Persons with sickle cell anemia or other hemoglobinopathies.
   * Persons with diseases requiring long-term aspirin therapy, such as rheumatoid arthritis or Kawasaki disease.
   * Persons with chronic renal dysfunction.
   * Persons with liver disorders.
   * Persons with active cancer.
   * Persons with chronic metabolic disease, such as diabetes mellitus, inherited metabolic disorders and mitochondrial disorders.
   * Persons with neuromuscular disorders, seizure disorders or cognitive dysfunction that may compromise the handling of respiratory secretions.
   * Residents of any age of nursing homes or other long-term care institutions.
   * Persons who are morbidly obese (Body Mass Index ≥40).
   * American Indians.
   * Alaskan natives.
2. Females of childbearing potential who are either pregnant, breast-feeding or are sexually active without the use of birth control. Female subjects of child-bearing potential that are sexually active must have a negative baseline pregnancy test and must agree to continue an acceptable method of birth control for the duration of the study and for 1 month post-treatment. A double barrier method, oral birth control pills administered for at least 2 monthly cycles prior to study drug administration, an intrauterine device (IUD), or medroxyprogesterone acetate administered intramuscularly for a minimum of one month prior to study drug administration are acceptable methods of birth control for inclusion into the study. Female subjects are considered of childbearing potential unless they are postmenopausal (absence of menstrual bleeding for 1 year - or 6 months if laboratory confirmation of hormonal status), or have had a hysterectomy, bilateral tubular ligation or bilateral ovariectomy.
3. Vaccination for seasonal influenza on or after August 1, 2015.
4. Receipt of any dose of nitazoxanide, oseltamivir, zanamivir, peramivir, amantadine or rimantadine within 30 days prior to screening.
5. Prior treatment with any investigational drug therapy within 30 days prior to screening.
6. Subjects with active respiratory allergies or subjects expected to require anti-allergy medications during the study period for respiratory allergies.
7. Known sensitivity to nitazoxanide or any of the excipients comprising the nitazoxanide tablets.
8. Subjects unable to take oral medications.
9. Subject has chronic kidney or liver disease (including Hepatitis A, B or C) or known impaired hepatic and/or renal function.
10. Presence of any other pre-existing chronic infection that is undergoing or requiring medical therapy.
11. Presence of any pre-existing illness that, in the opinion of the Investigator, would place the subject at an unreasonably increased risk through participation in this study.
12. Subjects who, in the judgment of the Investigator, will be unlikely to comply with the requirements of this protocol.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09-04 (Actual); Study Completion 2016-09-04 (Actual)

PRIMARY OUTCOMES:
Time to alleviation of all clinical symptoms of influenza | Up to 28 days

SECONDARY OUTCOMES:
Time to alleviation of each individual symptom of influenza | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Rossignol, M.D., Ph.D., Study Director — Romark Laboratories L.C.
Locations (27):
- United States (17):
  - Influence Study Site, Hot Springs, Arkansas
  - Influence Study Site, Anaheim, California
  - Influence Study Site, Fresno, California
  - Influence Study Site, Lomita, California
  - Influence Study Site, Kissimmee, Florida
  - Influence Study Site, Lauderdale Lakes, Florida
  - Influence Study Site, Saint Cloud, Florida
  - Influence Study Site, Columbus, Georgia
  - Influence Study Site, Savannah, Georgia
  - Influence Study Site, Lansdale, Pennsylvania
  - Influence Study Site, Rapid City, South Dakota
  - Influence Study Site, Jackson, Tennessee
  - Influence Study Site, Austin, Texas
  - Influence Study Site, Houston, Texas
  - Influence Study Site, Pharr, Texas
  - Influence Study Site, Plano, Texas
  - Influence Study Site, Waco, Texas
- Australia (9):
  - Influence Study Site, Brookvale, New South Wales
  - Influence Study Site, Castle Hill, New South Wales
  - Influence Study Site, Mosman, New South Wales
  - Influence Study Site, Browns Plains, Queensland
  - Influence Study Site, Springfield, Queensland
  - Influence Study Site, Berwick, Victoria
  - Influence Study Site, Lynbrook, Victoria
  - Influence Study Site, Rosebud, Victoria
  - Influence Study Site, Tarneit, Victoria
- Influence Study Site, San Juan, Puerto Rico